CLINICAL TRIAL: NCT05704543
Title: A Single-Dose Study to Evaluate the Relative Bioavailability, Safety, and Tolerability of SUBLOCADE at Alternative Injection Locations in Adults
Brief Title: Evaluation of Buprenorphine Extended-Release Subcutaneous Injection at Alternative Injection Locations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INDV-6000-405
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Opioid Use Disorder
Keywords: medicine for opioid use disorder (MOUD)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Extended-release Buprenorphine: Abdomen (Active Comparator): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the abdomen on Day 1.
  Interventions: Drug: Buprenorphine Extended-Release Injection
- Extended-release Buprenorphine: Upper Arm (Experimental): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the back of the upper arm on Day 1.
  Interventions: Drug: Buprenorphine Extended-Release Injection
- Extended-release Buprenorphine: Buttocks (Experimental): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the buttocks on Day 1.
  Interventions: Drug: Buprenorphine Extended-Release Injection
- Extended-release Buprenorphine: Thigh (Experimental): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the thigh on Day 1.
  Interventions: Drug: Buprenorphine Extended-Release Injection

INTERVENTIONS:
Drug: Buprenorphine Extended-Release Injection — Administered as a subcutaneous injection.
  Other Names: SUBLOCADE®

SUMMARY:
Extended-release buprenorphine (SUBLOCADE®) injection is currently approved for subcutaneous administration in the abdomen for treatment of opioid use disorder (OUD). Having alternative injection sites is desirable to provide additional flexibility to patients, particularly for those who may prefer less visible or more convenient injection locations.

The primary objective of this study is to assess the relative bioavailability of extended-release buprenorphine when administered at alternative injection locations (test treatments), in comparison to the abdomen (reference treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form (ICF) and have the ability to comply with the requirements and restrictions listed therein.
2. Sex: male or female.
3. Between the ages of 18 and 65 years inclusive, at the time of signing the ICF.
4. Currently meets Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for moderate or severe opioid use disorder (OUD), or documented history of moderate to severe OUD and receiving/stabilized on medicine for opioid use disorder (MOUD).
5. Body mass index: ≥ 18.0 to ≤ 33.0 kg/m^2.
6. New to treatment and seeking MOUD, or currently prescribed transmucosal (TM) buprenorphine (BUP) for OUD at the dose of 12 mg daily or can dose adjust to 12 mg daily.
7. Agree not to take any BUP-containing products, other than those administered for the current study, throughout the duration of the study.

Exclusion Criteria:

1. Has current diagnosis, other than OUD, requiring chronic opioid treatment.
2. Has concurrent primary substance use disorder, as defined by DSM-5 criteria, other than opioid, tobacco, cannabis, or mild to moderate alcohol use disorders.
3. Has target areas unsuitable for subcutaneous injections or evaluation of injections site (eg, nodules, scarring, lesions, excessive pigment) in the areas designated for possible injection in the study.
4. Has had significant traumatic injury or major surgical procedure (as defined by the investigator) within 30 days prior to the first dose of SUBLOCADE or still recovering from prior such injury or surgery.
5. Known personal and/or family history of congenital QT prolongation, or taking Class IA antiarrhythmic medications (eg, quinidine, procainamide, disopyramide) or Class III antiarrhythmic medications (eg, sotalol, amiodarone) or other medications that prolong the QT interval. Known family history of sudden unexplained death.
6. Currently taking (within the 30 days prior to signing the ICF) prescription or over-the-counter medications that are clinically relevant CYP 3A4 or CYP 2C8 inducers or inhibitors (eg, rifampin, azole antifungals [eg, ketoconazole], macrolide antibiotics [eg, erythromycin]).
7. Has history of suicidal ideation within 30 days prior to informed consent or history of a suicide attempt in the 6 months prior to informed consent.
8. Has any active medical condition, or psychiatric illness, or social/legal situation (including court order requiring treatment for OUD), or organ disease, or concurrent medication/treatment that may compromise participant safety, interfere with study endpoints, or limit compliance with study requirements, or compromise the ability of the participant to provide written informed consent.
9. Moderate or severe hepatic impairment (Child-Pugh B or C).
10. Has known allergy or hypersensitivity to BUP or any component of the ATRIGEL Delivery System.
11. Concurrent or has had prior treatment with any BUP long-acting injectable product (eg, SUBLOCADE) in the past 3 years prior to consent; or treatment with depot naltrexone within the 3 months prior to consent.
12. Treatment with another investigational agent within 30 days prior to Screening or enrollment in another clinical study (except for an observational study).
13. Concurrent treatment with medications contraindicated for use with BUP as per local prescribing information.
14. Is a member of site staff, has a financial interest in Indivior, or is an immediate family member of anyone directly involved in the study (ie, site staff or Indivior employee).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Director Clinical Development, Study Director — Indivior Inc.
Locations (6):
- United States (6):
  - Artemis Institute for Clinical Research, San Diego, California
  - Research Centers of America, Hollywood, Florida
  - Miami Lakes Medical Research, Miami Lakes, Florida
  - Rivus Wellness and Research Institute, Oklahoma City, Oklahoma
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laffont CM, Lapeyra O, Mangal D, Dobbins R. A Single-Dose Study to Evaluate the Relative Bioavailability, Safety, and Tolerability of Monthly Extended-Release Buprenorphine at Alternative Injection Locations in Adult Participants with Opioid Use Disorder. Clin Drug Investig. 2024 Dec;44(12):939-949. doi: 10.1007/s40261-024-01406-7. Epub 2024 Nov 14. PMID 39543001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 175 participants were screened to assess eligibility; of these, 132 received SUBOXONE during the Run-In Period (all eligible participants were attempted to be stabilized on 12 mg SUBOXONE [buprenorphine/naloxone] sublingual film once daily for a minimum of 7 days before the SUBLOCADE injection). 44 participants discontinued during the Run-In Period. A total of 88 participants were thus randomized (Started) to a treatment arm to receive extended-release buprenorphine on Day 1.
Period: Overall Study
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Started | 22 | 21 | 22 | 23
Completed | 20 | 18 | 22 | 21
Not Completed | 2 | 3 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh | Total
Number analyzed (Participants) | 22 | 21 | 22 | 23 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (10.35) | 43.9 (9.61) | 45.6 (8.94) | 36.7 (7.89) | 41.2 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 11 | 31
  Male | 15 | 15 | 15 | 12 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 5 | 15
  Not Hispanic or Latino | 19 | 17 | 19 | 18 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 8 | 4 | 25
  White | 14 | 14 | 13 | 18 | 59
  More than one race | 1 | 0 | 1 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 22 | 23 | 88
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.87 (4.698) | 25.95 (5.011) | 26.06 (4.259) | 26.30 (4.500) | 26.30 (4.552)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Study Day 1 to Day 29 (AUC0-28days) of Buprenorphine
Time Frame: Day 1 at predose and at 1, 2, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48 hours post-dose and on Days 4, 6, 8, 11, 15, 18, 22, 25, and 29
Population: Pharmacokinetic Evaluable Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Number analyzed (Participants) | 22 | 17 | 22 | 21
h*ng/mL | 1640 (41.8) | 1720 (57.4) | 1570 (42.7) | 1870 (56.2)

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Buprenorphine
Time Frame: as for outcome 1
Population: Pharmacokinetic Evaluable Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Number analyzed (Participants) | 22 | 20 | 22 | 21
ng/mL | 6.61 (46.9) | 9.17 (85.8) | 7.11 (39.7) | 10.1 (73.2)

3. Secondary Outcome: Participants With Treatment-emergent Adverse Events
Time Frame: 28 days
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Number analyzed (Participants) | 22 | 21 | 22 | 23
Percentage of participants
  Any treatment-emergent adverse event (TEAE) | 22.7 | 14.3 | 18.2 | 8.7
  TEAE identified as injection site reaction | 9.1 | 4.8 | 4.5 | 4.3
  Related TEAE | 9.1 | 4.8 | 13.6 | 4.3
  Severe TEAE | 0 | 0 | 0 | 0
  TEAE of opioid withdrawal symptom | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Identified as Injection Site Reactions
Time Frame: 28 days
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Number analyzed (Participants) | 22 | 21 | 22 | 23
Percentage of participants
  Injection site erythema | 4.5 | 0 | 4.5 | 0
  Injection site induration | 0 | 4.8 | 4.5 | 0
  Injection site pain | 4.5 | 4.8 | 0 | 0
  Injection site swelling | 0 | 4.8 | 0 | 4.3
  Injection site reaction | 4.5 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events
Time Frame: 28 days
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Number analyzed (Participants) | 22 | 21 | 22 | 23
Percentage of participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Injection Site Grading
Description: Injection sites will be assessed for pain, tenderness, erythema/redness, induration, or swelling. Local injection site tolerability will be assigned a severity grade, including none (grade 0), mild (grade 1), moderate (grade 2), severe (grade 3), or potentially life-threatening (grade 4) utilizing the Injection Site Grading Scale.
Time Frame: Day 1 at 10 minutes and 2 hours post dosing
Population: Safety Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Number analyzed (Participants) | 22 | 21 | 22 | 23
Percentage of participants
  Pain, None (Grade 0) at 10 minutes | 59.1 | 57.1 | 68.2 | 56.5
  Pain, Mild (Grade 1) at 10 minutes | 31.8 | 28.6 | 18.2 | 34.8
  Pain, Moderate (Grade 2) at 10 minutes | 9.1 | 14.3 | 13.6 | 8.7
  Tenderness, None (Grade 0) at 10 minutes | 59.1 | 66.7 | 77.3 | 56.5
  Tenderness, Mild (Grade 1) at 10 minutes | 31.8 | 33.3 | 22.7 | 39.1
  Tenderness, Moderate (Grade 2) at 10 minutes | 9.1 | 0 | 0 | 4.3
  Erythema/redness, None (Grade 0) at 10 minutes | 86.4 | 81.0 | 86.4 | 100.0
  Erythema/redness, Mild (Grade 1) at 10 minutes | 13.6 | 19.0 | 13.6 | 0
  Induration, None (Grade 0) at 10 minutes | 95.5 | 85.7 | 95.5 | 87.0
  Induration, Mild (Grade 1) at 10 minutes | 4.5 | 14.3 | 4.5 | 13.0
  Injection site swelling, None (Grade 0) at 10 minutes | 90.9 | 85.7 | 90.9 | 82.6
  Injection site swelling, Mild (Grade 1) at 10 minutes | 9.1 | 14.3 | 9.1 | 17.4
  Pain, None (Grade 0) at 2 hours | 100.0 | 81.0 | 90.9 | 91.3
  Pain, Mild (Grade 1) at 2 hours | 0 | 19.0 | 9.1 | 8.7
  Tenderness, None (Grade 0) at 2 hours | 86.4 | 81.0 | 95.5 | 91.3
  Tenderness, Mild (Grade 1) at 2 hours | 13.6 | 19.0 | 4.5 | 8.7
  Erythema/redness, None (Grade 0) at 2 hours | 95.5 | 90.5 | 95.5 | 100.0
  Erythema/redness, Mild (Grade 1) at 2 hours | 4.5 | 9.5 | 4.5 | 0
  Induration, None (Grade 0) at 2 hours | 86.4 | 81.0 | 95.5 | 95.7
  Induration, Mild (Grade 1) at 2 hours | 13.6 | 19.0 | 4.5 | 4.3
  Injection site swelling, None (Grade 0) at 2 hours | 95.5 | 85.7 | 90.9 | 87.0
  Injection site swelling, Mild (Grade 1) at 2 hours | 4.5 | 14.3 | 9.1 | 13.0

7. Secondary Outcome: Injection Site Pain
Description: Measured on a 100 mm visual analog scale (VAS), where 0 represents no pain and 100 represents maximum pain.
Time Frame: Day 1 at 1, 5, 10, 15, and 30 minutes post dosing
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extended-release Buprenorphine: Abdomen | Extended-release Buprenorphine: Upper Arm | Extended-release Buprenorphine: Buttocks | Extended-release Buprenorphine: Thigh
Number analyzed (Participants) | 22 | 21 | 22 | 23
score on a scale
  1 minute | 37.5 (27.95) | 29.0 (24.10) | 27.4 (32.02) | 29.3 (28.99)
  5 minutes | 23.2 (26.13) | 16.0 (16.59) | 13.6 (23.62) | 19.0 (23.56)
  10 minutes | 12.0 (14.88) | 9.4 (11.80) | 8.2 (14.15) | 12.5 (21.30)
  15 minutes | 4.8 (6.58) | 6.0 (8.76) | 4.9 (11.80) | 8.6 (20.64)
  30 minutes | 1.8 (2.56) | 4.5 (8.69) | 1.4 (2.46) | 6.6 (19.93)

ADVERSE EVENTS:
Time Frame: Up to 86 days
Groups:
- Pre-injection (Run-In Period): Participants who received SUBOXONE during the Run-In Period (all eligible participants were attempted to be stabilized on 12 mg SUBOXONE [buprenorphine/naloxone] sublingual film once daily for a minimum of 7 days before injection with extended-release buprenorphine). 44 participants discontinued during the Run-In Period.
- Extended-release Buprenorphine: Abdomen (Post-injection): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the abdomen on Day 1.
  Buprenorphine Extended-Release Injection: Administered as a subcutaneous injection.
- Extended-release Buprenorphine: Upper Arm (Post-injection): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the back of the upper arm on Day 1.
  Buprenorphine Extended-Release Injection: Administered as a subcutaneous injection.
- Extended-release Buprenorphine: Buttocks (Post-injection): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the buttocks on Day 1.
  Buprenorphine Extended-Release Injection: Administered as a subcutaneous injection.
- Extended-release Buprenorphine: Thigh (Post-injection): Participants will receive a single, subcutaneous injection of 300 mg extended-release buprenorphine in the thigh on Day 1.
  Buprenorphine Extended-Release Injection: Administered as a subcutaneous injection.
Arm/Group | Pre-injection (Run-In Period) | Extended-release Buprenorphine: Abdomen (Post-injection) | Extended-release Buprenorphine: Upper Arm (Post-injection) | Extended-release Buprenorphine: Buttocks (Post-injection) | Extended-release Buprenorphine: Thigh (Post-injection)
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/22 | 0/21 | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/22 | 0/21 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 26/132 | 5/22 | 3/21 | 4/22 | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-injection (Run-In Period) (N=132) | Extended-release Buprenorphine: Abdomen (Post-injection) (N=22) | Extended-release Buprenorphine: Upper Arm (Post-injection) (N=21) | Extended-release Buprenorphine: Buttocks (Post-injection) (N=22) | Extended-release Buprenorphine: Thigh (Post-injection) (N=23)
General disorders and administration site conditions (General disorders) | 2 | 2 | 2 | 1 | 1
Gastrointestinal disorders (Gastrointestinal disorders) | 14 | 0 | 1 | 1 | 0
Infections and infestations (Infections and infestations) | 4 | 2 | 0 | 0 | 0
Investigations (Investigations) | 1 | 0 | 0 | 1 | 1
Immune system disorders (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Nervous system disorders (Nervous system disorders) | 6 | 1 | 0 | 0 | 0
Psychiatric disorders (Psychiatric disorders) | 6 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT05704543/Prot_000.pdf
  • Statistical Analysis Plan: Primary (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT05704543/SAP_001.pdf
  • Statistical Analysis Plan: Addendum (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT05704543/SAP_002.pdf